CLINICAL TRIAL: NCT05154318
Title: Study Comparing the Efficacy of Pericapsular Nerve Group (PENG) Block and Facia Iliaca Compartment Block (FICB) in Hip Fracture - A Prospective Randomised Controlled Trial
Brief Title: Efficacy of Pericapsular Nerve Group Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Dr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW21-382
Record Dates: First submitted 2021-11-29; First posted 2021-12-13 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular Nerve Group Block (Experimental): 30ml 0.3% Ropivacaine will be injected between psoas muscle and iliopubic eminence.
  Interventions: Procedure: Pericapsular Nerve Group Block
- Fascia iliaca compartment block (Active Comparator): 30ml 0.3% Ropivacaine will be injected into fascia iliaca compartment.
  Interventions: Procedure: Fascia iliaca compartment block

INTERVENTIONS:
Procedure: Pericapsular Nerve Group Block — Nerve block targeting major hip joint sensory nerves.
  Arms: Pericapsular Nerve Group Block
Procedure: Fascia iliaca compartment block — Routine nerve block for hip fracture surgery.
  Arms: Fascia iliaca compartment block

SUMMARY:
Hip fracture is a common orthpaedic problem especially in elderly population. Fascia iliaca compartment block (FICB) and femoral nerve block are well-established technique as part of peri-operative multimodal analgesia for hip fractures. Reviews have shown peripheral nerve blocks including FICB, femoral nerve block and 3-in-1 block could reduce both pain and opioid consumption compared with systematic analgesia. However, there are also literature suggesting that some nerves that account for the major hip joint sensory innervation are not consistently covered. As a result, a new ultrasound guided regional technique, Pericapsular Nerve Group Block (PENG) was introduced in 2018. The primary aim of this study is to compare the analgesic effect of PENG block and FICB in terms of pain score during post-operative period. It also compares the range of movement, quadriceps power and other parameters related to physical functions of the operated hip as secondary outcomes.

DETAILED DESCRIPTION:
Hip fracture is a common orthopaedic problem especially in elderly population. The number of hip fractures each year is expected to double from 2.2 million in 2017 to 4.5 million in 2050. It is the commonest reason for elderly to require hospitalisation and emergency operation. Significant morbidities such as pulmonary embolism, pneumonia and bed sore can be resulted from immobility and pain. Hip fracture also contributes to post-operative mortality at a rate about 8% at 1 month and 30% at 1 year.

Fascia iliaca compartment block (FICB) and femoral nerve block are well-established technique as part of peri-operative multimodal analgesia for hip fractures. Cochrane review has shown peripheral nerve blocks including FICB, Femoral nerve block and 3-in-1 block could reduce both pain at 30 minute and opioid consumption compared with systemic analgesia. In particular, FICB is found to be superior to opioids for pain control on movement, preoperative analgesic consumption, time to first analgesic request, and time to perform spinal anaesthesia. However, literature suggests that the obturator nerve is not consistently covered.

The anterior hip capsule which contributes the major hip joint sensory innervation is supplied by femoral nerve (FN), obturator nerve (ON) and accessory obturator nerve (AON). As a result, a novel ultrasound guided regional technique, Pericapsular Nerve Group Block (PENG) was introduced in 2018, targeting the above 3 nerves. This is very important as the obturator nerve is also blocked with this technique. Case reports showed reduction in pain scores compared with baseline 30 minutes after block placement and no clinically evident quadriceps weakness was detected.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Age 18 or above
* Scheduled for hip fracture corrective surgery in Queen Mary Hospital
* Chinese patients
* Able to provide informed oral and written consent
* Abbreviated Mental Test (AMT) 7 or above

Exclusion Criteria:

* Patient refusal
* ASA III or above
* Allergy to local anaesthetics, opioids, paracetamol, NSAID including COX-2 inhibitors
* Operation delayed for more than 2 days on admission
* Pre-existing peripheral neuropathy or history of stroke
* Preoperative non-walker
* Pre-existing osteoarthritis of knee (KL grade 4)
* Multiple fractures (additional to hip fracture)
* Sepsis
* Impaired renal function (Defined as preoperative creatinine level >120 μmol or eGFR <50% of normal reference for their age group
* Patient with coagulopathy (Platelet < 100 or INR >1.5)
* Prior surgery at the inguinal or supra-inguinal area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score at rest on postoperative day 1 | on postoperative day 1
  Measure pain score at rest using numerical rating scale from 0 to 10, where 0 is no pain and 10 is the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Timmy CW Chan, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Timmy Chan, Hong Kong, Hong Kong